CLINICAL TRIAL: NCT05031507
Title: Clinical and Laboratory Study of Rare Skeletal Disorders
Brief Title: Study of Skeletal Disorders
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000213; 000213-CH
Record Dates: First submitted 2021-09-01; First posted 2021-09-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Skeletal Disorders
Keywords: skeletal; Bone; Skeletal Dysplasia; Short Stature; DWARFISM; Natural History
MeSH Terms: conditions — Mucopolysaccharidosis IV; Dwarfism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Subjects with rare skeletal disorders

SUMMARY:
Background:

There are 461 conditions that affect the bones (skeletal disorders). Many of these are not well understood and do not have any specific treatments. Researchers want to collect more data about these conditions.

Objective:

To gain more information about the causes of skeletal disorders and how they progress over time.

Eligibility:

People ages 2 months or older with known or suspected skeletal disorders or history of pregnancy affected by skeletal findings. Also, healthy family members of affected enrolled participants.

Design:

Participants can take part in the study either remotely or in person. Those who take part remotely may send in medical records, blood samples, photographs, and other materials.

Participants medical records will be reviewed. They may give blood and/or urine samples. They will give blood, saliva, or tissue samples for genetic tests. They may have genetic counseling.

Participants ages 2 years and older may have different kinds of imaging scans, such as x-rays. For these scans, they may have to lie still while machines take pictures of their bones.

Participants with skeletal disorders who come to the clinic will be examined. They may be asked to stay in the hospital for a few days to take extra tests. They may have a bone or skin biopsy.

Participants with skeletal disorders may be photographed to show the effects of their disorder and how it changes over time.

For participants with skeletal disorders, their blood or tissue samples may be used to make a special type of stem cell. These cells can be used in the laboratory to make many other types of cells. A large supply of these cells may be created for research.

Participation will last indefinitely.

DETAILED DESCRIPTION:
Study Description:

This is a clinical and laboratory study of rare skeletal disorders using a combination of both retrospective and prospective methods. This is a single site study taking place at the NIH Clinical Center with the added ability for participants to submit medical records and specimens remotely.

Objectives:

Primary Objective: To provide a protocol in which subjects with rare skeletal disorders can be evaluated and studied and to allow for the receipt of tissues and clinical specimens from individuals and investigators outside of the NIH

Secondary Objective: To perform genetic testing including genes currently known to cause skeletal disorders as well as those currently without association with skeletal disorders

Endpoints:

Primary Endpoint: To define or further define genetic etiologies of known and unknown skeletal disorders and create genotype-phenotype correlations when possible

Secondary Endpoints: To describe natural history of individual disorders if enough data is collected on a particular condition(s)

ELIGIBILITY:
* INCLUSION CRITERIA:

Our study population will support the mission and scientific focus of the Unit on Skeletal Genomics. We will focus enrollment of subjects (and their relatives) who fall within one of the below categories:

* Individuals with a skeletal disorder that affects phosphate levels and/or metabolism
* Individuals with a skeletal disorder associated with skeletal overgrowth
* Individuals with a skeletal disorder or history of pregnancy affected by skeletal findings with an unknown molecular basis or unknown etiology

In addition to noting the above, to be eligible to participate in this study as an affected subject, an individual must meet all of the following criteria:

1. Have a known (via clinical, radiographic or molecular diagnosis) or suspected skeletal disorder, findings associated with or increasing risk for skeletal abnormalities, or history of pregnancy affected by skeletal findings
2. State willingness to comply with study procedures and availability for the duration of the study
3. Be age 2 months or older
4. Be able to understand and sign informed consent document (or availability of a parent/guardian or LAR to provide written consent)

In order to be eligible to participate in this study as an unaffected subject, an individual must meet all of the following criteria:

1. Be an unaffected family member of an affected enrolled subject
2. State willingness to comply with study procedures and availability for the duration of the study
3. Be age 2 months or older
4. Be able to understand and sign informed consent document (or availability of a parent/guardian)

EXCLUSION CRITERIA:

The below describe exclusion criteria for an individual to participate as an affected subject:

1. An individual who cannot or is unwilling to abide by the procedures of the protocol.
2. An individual deemed to not have sufficient signs of or risks for skeletal disease.
3. An individual who is pregnant.

The below describe exclusion criteria for an individual to participate as an unaffected subject:

1. An individual who cannot or is unwilling to abide by the procedures of the protocol.
2. An individual that shows signs of skeletal disease.
3. An individual who is pregnant.

Ages: 2 Months to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study cohort will include individuals with known (via clinical, radiographic or molecular diagnosis) or suspected skeletal disorders, findings associated with or increasing risk for skeletal abnormalities, or history of pregnancy affected by skeletal findings.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
To define or further define genetic etiologies of known and unknown skeletal disorders and create genotype-phenotype correlations when possible | ongoing
  To define or further define genetic etiologies of known and unknown skeletal disorders and create genotype-phenotype correlations when possible

SECONDARY OUTCOMES:
Describe Natural History | ongoing
  To describe natural history of individual disorders if enough data is collected on a particular condition(s)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos R Ferreira Lopez, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000213-CH.html